CLINICAL TRIAL: NCT02329548
Title: Qualitative Sweat Distribution Among Youth With Postural Tachycardia Syndrome (POTS), Syncope, or Anxiety
Brief Title: Qualitative Sweat Distribution During Tilt Table Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Geoffrey Heyer, Assistant Professor of Neurology and Pediatrics, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB14-00528
Record Dates: First submitted 2014-12-12; First posted 2014-12-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Postural Tachycardia Syndrome; Syncope; Anxiety
Keywords: Alizarin; Orthostatic; POTS; Tilt table testing; Syncope; Anxiety
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Syncope; Anxiety Disorders | interventions — alizarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alizarin Red (Experimental): All participating patients will undergo the Alizarin Red intervention.
  Interventions: Other: Alizarin Red

INTERVENTIONS:
Other: Alizarin Red — An Alizarin Red mixture will be applied to all exposed skin below the angle of the mandible. Once applied the patient will be tilted to 70 degrees. Serial photos will be taken once sweat begins and until conclusion of the test.

SUMMARY:
This study uses an Alizarin Red powder mixture to characterize the sweat distributions in youth during tilt table testing. Patients with a known orthostatic sweat response from a prior clinical tilt table test in the investigators laboratory will be recruited. The Alizarin Red powder will be applied to exposed skin, and quantitative sweat will be measured at the thigh. During tilt testing, serial photos will be taken once the sweat response occurs. Sweat distributions will be compared during syncope (orthostatic sweat), during periods of anxiety (emotional sweat), and in patients with POTS (with and without syncope).

DETAILED DESCRIPTION:
The investigators' laboratory has conducted an exploratory study of quantitative sweat during tilt table testing over the past year. Some patients with Postural Tachycardia Syndrome (POTS) experience excessive sweating. Patients with syncope (without POTS) have an increase in sweat during their tilt-induced syncopal episode. Increased warmth and sweating can be among the first pre-syncopal symptoms in some individuals. Anxiety can also produce a sweat response, so-called "emotional sweating". Emotional sweating tends to affect the palms, soles, and forehead prominently, while the distribution of orthostatic sweat has not been well-described. The investigators' sweat measure quantifies sweat production, but placement of the sweat capsules is limited to four sites on the arms and legs.

An Alizarin Red powder mixture applied to exposed skin is brown in color when dry and red in color when moist. Using Alizarin red, a quantitative sweat measure, and serial photography, the investigators will characterize the sweat distribution in patients with syncope, anxiety, and POTS. Patients will be recruited if they had a sweat response from prior tilt table testing performed in the investigators' laboratory.

Consenting patients will wear underwear or bathing suits. The investigators will apply Alizarin Red to all exposed skin below the angle of the mandible. A single sweat capsule will be placed at the right hip. Pre-tilt photos will be taken, and then the patient will be tilted head-upright to seventy degrees. Once sweat begins, serial photos will be taken. The patient will remain in the tilted position until syncope occurs or the Alizarin powder is saturated red. If a sweat response is not prominent and syncope does not occur, the patient will be lowered after 30 minutes. The investigators will use the serial photos to describe the temporal distribution of sweat with each patient.

Orthostatic sweat can occur before or after syncope, but based on the investigators' prior quantitative sweat measures, there is always an associated drop in blood pressure. The investigators can distinguish emotional from orthostatic sweat based on the patient's self-report of anxiety/panic, the presence of tachypnea, and the absence of syncope or hypotension.

The current study aims to characterize sweat production during tilt testing and distinguish orthostatic and emotional sweat distributions. The primary goal of this study is to compare sweat distributions in patients during syncope (orthostatic sweat) and during anxiety (emotional sweat). The secondary goal is to characterize tilt-induced sweat distributions in POTS patients and compare them to the orthostatic and emotional sweat patterns. The investigators hypothesize that emotional sweat will predominantly affect the palms and soles (forehead sweat will not be measured), while orthostatic sweat will have a truncal predominance. This study is significant because the sweat pattern may help to resolve POTS and syncope phenotypes which will ultimately aid in gene discovery for these disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Must have prior documented sweat response from tilt table testing in our laboratory.
2. Must speak English well enough to describe orthostatic symptoms and imminent syncope.

Exclusion Criteria:

1. Pregnancy
2. Somatic or psychiatric illness that precludes tilt table testing
3. Skin defect or rash that precludes application of Alizarin Red powder
4. Known sweat disorder of any type
5. Long QT syndrome

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Orthostatic versus emotional sweat distribution assessed by serial photography | Up to 30 minutes
  The temporal and regional sweat distributions will be assessed by serial photography. Orthostatic sweat will be distinguished from emotional sweat based on the presence of hypotension/syncope, self-report of anxiety, and presence of tachypnea (emotional sweat).

SECONDARY OUTCOMES:
Sweat distribution among patients with POTS assessed by serial photography | Up to 30 minutes
  Using serial photography the temporal and regional distribution of sweat among POTS patients will be compared to syncope-only patients and patients with anxiety (without hypotension).

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey L. Heyer, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, neurology outpatient clinic, Columbus, Ohio, United States